CLINICAL TRIAL: NCT05067881
Title: Post COVID-19 Pneumo-hematocele: Clinical Presentation and Treatment Pathway
Brief Title: Post-COVID-19 Pneumo-hematocele
Acronym: PHC
Status: Completed | Type: Observational
Sponsor: Hospital General Ajusco Medio (Other)
Collaborators: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Karla Verónica Chavez-Tostado, Head of Surgery department, Hospital General Ajusco Medio
Other Study IDs: HGAM02
Record Dates: First submitted 2021-09-28; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Respiratory Infection
Keywords: COVID-19; Pneumohematocele; Giant bullae; Pneumatocele
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pneumohematocele: Patients with SARS CoV-2 diagnosis and PHC on imaging studies
  Interventions: Procedure: Pulmonary resection

INTERVENTIONS:
Procedure: Pulmonary resection — Resection of pneumohematocele

SUMMARY:
Introduction. As the COVID-19 pandemic has continued, an increasing number of long-term complications are emerging. Recently, the appearance of characteristic pulmonary lesions has been noted, being described as post COVID-19 pneumatocele. The aim of this study is to describe the clinical, histopathologic and imaging features of post COVID-19 pneumo-hematoceles (PHC) and secondarily to suggest a treatment algorithm in these patients.

Methods. A retrospective study was performed in patients admitted with diagnosis of SARS-CoV2 infection from March 2020 to September 2021 who presented PHC on imaging studies. Clinical and demographic variables were recorded and CT scans were analyzed. A logistic regression analysis was performed to determine the risk for rupture according to PHC characteristics.

It appears that PHC occurs secondary to encapsulation of blood accumulation, the result of micro capillary bleeding, with partial reabsorption of blood and subsequent air filling. The recommendation is to operate on patients with PHC of 5cm and those with persistent lesions of 3cm.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a positive protein chain reaction for SARS-CoV2,
* PHC on imaging studies.

Exclusion Criteria:

* loss of follow up
* age out of range.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a positive chain reaction for SARS CoV-2 who had PHC on imaging studies in two hospitals of Mexico City
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
PHC diagnosis | From date of diagnosis until 4 weeks after diagnosis
  Pneumohematoceles on imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: Karla V Chavez Tostado, MD, Principal Investigator — Head of surgery department
Locations (1):
- Karla Verónica Chávez Tostado, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ho JS, Sia CH, Chan MY, Lin W, Wong RC. Coronavirus-induced myocarditis: A meta-summary of cases. Heart Lung. 2020 Nov-Dec;49(6):681-685. doi: 10.1016/j.hrtlng.2020.08.013. Epub 2020 Aug 20. PMID 32861884
- [Background] Inciardi RM, Lupi L, Zaccone G, Italia L, Raffo M, Tomasoni D, Cani DS, Cerini M, Farina D, Gavazzi E, Maroldi R, Adamo M, Ammirati E, Sinagra G, Lombardi CM, Metra M. Cardiac Involvement in a Patient With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):819-824. doi: 10.1001/jamacardio.2020.1096. PMID 32219357
- [Background] Chen X, Laurent S, Onur OA, Kleineberg NN, Fink GR, Schweitzer F, Warnke C. A systematic review of neurological symptoms and complications of COVID-19. J Neurol. 2021 Feb;268(2):392-402. doi: 10.1007/s00415-020-10067-3. Epub 2020 Jul 20. PMID 32691236
- [Background] Maury A, Lyoubi A, Peiffer-Smadja N, de Broucker T, Meppiel E. Neurological manifestations associated with SARS-CoV-2 and other coronaviruses: A narrative review for clinicians. Rev Neurol (Paris). 2021 Jan-Feb;177(1-2):51-64. doi: 10.1016/j.neurol.2020.10.001. Epub 2020 Dec 16. PMID 33446327
- [Background] Ojo AS, Balogun SA, Williams OT, Ojo OS. Pulmonary Fibrosis in COVID-19 Survivors: Predictive Factors and Risk Reduction Strategies. Pulm Med. 2020 Aug 10;2020:6175964. doi: 10.1155/2020/6175964. eCollection 2020. PMID 32850151
- [Background] Gentile F, Aimo A, Forfori F, Catapano G, Clemente A, Cademartiri F, Emdin M, Giannoni A. COVID-19 and risk of pulmonary fibrosis: the importance of planning ahead. Eur J Prev Cardiol. 2020 Sep;27(13):1442-1446. doi: 10.1177/2047487320932695. Epub 2020 Jun 17. No abstract available. PMID 32551971
- [Background] Sun R, Liu H, Wang X. Mediastinal Emphysema, Giant Bulla, and Pneumothorax Developed during the Course of COVID-19 Pneumonia. Korean J Radiol. 2020 May;21(5):541-544. doi: 10.3348/kjr.2020.0180. Epub 2020 Mar 20. PMID 32207255
- [Background] Sato L, Kinoshita N, Nakamoto T, Ohmagari N. Hemoptysis and a Newly Formed Lung Bulla in a Case of Convalescent COVID-19 Pneumonia. Intern Med. 2021 Mar 1;60(5):803-805. doi: 10.2169/internalmedicine.5684-20. Epub 2021 Jan 15. PMID 33456035
- [Background] Xu W, Luo X, Wang H, Shen C, Song Y, Sun T, Chen M. Pulmonary emphysema, bullae, and pneumothorax in COVID-19 pneumonia. Radiol Case Rep. 2021 May;16(5):995-998. doi: 10.1016/j.radcr.2021.01.055. Epub 2021 Jan 31. PMID 33552325
- [Background] Sanivarapu RR, Farraj K, Sayedy N, Anjum F. Rapidly developing large pneumatocele and spontaneous pneumothorax in SARS-CoV-2 infection. Respir Med Case Rep. 2020;31:101303. doi: 10.1016/j.rmcr.2020.101303. Epub 2020 Dec 2. PMID 33294361
- [Background] Hamad AM, El-Saka HA. Post COVID-19 large pneumatocele: clinical and pathological perspectives. Interact Cardiovasc Thorac Surg. 2021 Jul 26;33(2):322-324. doi: 10.1093/icvts/ivab072. PMID 33764376
- [Background] Sharma S, Kasi A. Pneumatocele. 2025 Jan 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK556146/ PMID 32310606
- [Background] Desrues B, Delaval P, Motreff C, Kernec J, Dormoy C, Pencole C, Bergeron D, Malledan Y, Saint-Marc C. [Post-traumatic pneumatocele and hemato-pneumatocele of the lung. Apropos of 3 cases]. Rev Mal Respir. 1988;5(1):67-70. French. PMID 3368637
- [Background] Kaira K, Ishizuka T, Yanagitani N, Sunaga N, Hisada T, Mori M. Pulmonary traumatic pneumatocele and hematoma. Jpn J Radiol. 2009 Feb;27(2):100-2. doi: 10.1007/s11604-008-0296-x. Epub 2009 Mar 12. PMID 19373539
- [Background] Al-Ghafri M, Al-Hanshi S, Al-Ismaily S. Two Cases of Pneumatoceles in Mechanically Ventilated Infants. Oman Med J. 2015 Jul;30(4):299-302. doi: 10.5001/omj.2015.59. PMID 26366266
- [Background] Liu K, Zeng Y, Xie P, Ye X, Xu G, Liu J, Wang H, Qian J. COVID-19 with cystic features on computed tomography: A case report. Medicine (Baltimore). 2020 May;99(18):e20175. doi: 10.1097/MD.0000000000020175. PMID 32358406
- [Background] Purdy GD, Cullen M, Yedlin S, Bedard MP. An unusual neonatal case presentation: Streptococcus pneumoniae pneumonia with abscess and pneumatocele formation. J Perinatol. 1987 Fall;7(4):378-81. No abstract available. PMID 3333168
- [Background] Ishiguchi S, Nishioka K, Kanetake Y, Sugiyama K, Shibayama M. [Pneumatocele accompanying staphylococcal pneumonia]. Rinsho Hoshasen. 1966 Aug;11(8):644-53. No abstract available. Japanese. PMID 5182446
- [Background] Sandhu JS, Goodman PC. Pulmonary cysts associated with Pneumocystis carinii pneumonia in patients with AIDS. Radiology. 1989 Oct;173(1):33-5. doi: 10.1148/radiology.173.1.2789413.
- [Background] Murayama D, Kojima D, Hino A, Yamamoto Y, Doiuchi T, Horikawa A, Kurihara H. A case of bulla formation after treatment for COVID-19 pneumonia. Radiol Case Rep. 2021 May;16(5):1162-1164. doi: 10.1016/j.radcr.2021.03.003. Epub 2021 Mar 10. PMID 33728014
- [Background] Capleton P, Ricketts W, Lau K, Ellis S, Sheaff M, Giaslakiotis K, Uys S, Tchrakian N. Pneumothorax and Pneumatocoele Formation in a Patient with COVID-19: a Case Report. SN Compr Clin Med. 2021;3(1):269-272. doi: 10.1007/s42399-020-00689-z. Epub 2021 Jan 7. PMID 33432305
- [Background] Hansell DM, Bankier AA, MacMahon H, McLoud TC, Muller NL, Remy J. Fleischner Society: glossary of terms for thoracic imaging. Radiology. 2008 Mar;246(3):697-722. doi: 10.1148/radiol.2462070712. Epub 2008 Jan 14. PMID 18195376
- [Background] Fan Q, Pan F, Yang L. Spontaneous pneumothorax and subpleural bullae in a patient with COVID-19: a 92-day observation. Eur J Cardiothorac Surg. 2020 Oct 1;58(4):858-860. doi: 10.1093/ejcts/ezaa305. PMID 32951046
- [Background] Wu J, Feng LC, Xian XY, Qiang J, Zhang J, Mao QX, Kong SF, Chen YC, Pan JP. [Novel coronavirus pneumonia (COVID-19) CT distribution and sign features]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Apr 12;43(4):321-326. doi: 10.3760/cma.j.cn112147-20200217-00106. Chinese. PMID 32125131
- [Background] Bernheim A, Mei X, Huang M, Yang Y, Fayad ZA, Zhang N, Diao K, Lin B, Zhu X, Li K, Li S, Shan H, Jacobi A, Chung M. Chest CT Findings in Coronavirus Disease-19 (COVID-19): Relationship to Duration of Infection. Radiology. 2020 Jun;295(3):200463. doi: 10.1148/radiol.2020200463. Epub 2020 Feb 20. PMID 32077789
- [Derived] Chavez KV, Pimienta-Ibarra AS, Maruquez-Gonzalez H, Flores-Garces JC, Pena-Mirabal ES, Bolanos-Morales FV. Post COVID-19 pneumo-hematocele: clinical presentation and treatment pathway. Gen Thorac Cardiovasc Surg. 2022 Jun;70(6):566-574. doi: 10.1007/s11748-022-01771-0. Epub 2022 Jan 18. PMID 35041128